CLINICAL TRIAL: NCT01459861
Title: Assessment of Early Ambulation in Patients Receiving Continuous Adductor Canal Block With Ultrasound Guided Posterior Capsular Knee Injection vs. Femoral Nerve Block With Tibial Nerve Block Following Total Knee Replacement
Brief Title: Early Ambulation After Adductor Canal Block for Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively closed early
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-09-003
Record Dates: First submitted 2011-10-06; First posted 2011-10-26 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-02

CONDITIONS: Pain; Osteoarthritis
Keywords: early ambulation; knee arthroplasty
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canal Block and Capsular Injection (Experimental): Adductor canal block with a continuous catheter and ultrasound guided posterior capsular injection with local anesthetic solution.
  Interventions: Procedure: Canal Block and Capsular Injection
- Femoral with Tibial Nerve Block (Active Comparator): Continuous femoral nerve block with catheter and selective tibial nerve block in the popliteal fossa.
  Interventions: Procedure: Femoral Nerve Block with Tibial Nerve Block

INTERVENTIONS:
Procedure: Canal Block and Capsular Injection — Continuous Adductor canal block with 15ml of ropivacaine 0.2% with epinephrine 1:400,000 followed by an infusion of ropivacaine 0.2% at 6ml per hour for 2 days post operatively. This is combined with ultrasound guided posterior capsular knee injection with 30ml ropivacaine 0.2% with epinephrine 1:400,000.
  Arms: Canal Block and Capsular Injection
Procedure: Femoral Nerve Block with Tibial Nerve Block — Continuous femoral nerve block with 15ml of ropivacaine 0.2% followed by an infusion of ropivacaine 0.2% at 6ml per hour for 2 days after surgery combined with tibial nerve block in the popliteal fossa with ropivacaine 0.5% up to 15ml.
  Arms: Femoral with Tibial Nerve Block

SUMMARY:
The purpose of this study is to assess early ambulation following total knee replacement in patients receiving continuous adductor canal block with posterior capsular injection compared to continuous femoral nerve block with tibial nerve block.

ELIGIBILITY:
Inclusion Criteria:

* knee arthroplasty
* ages 18-80

Exclusion Criteria:

* history of neurological disease
* diabetes
* pregnancy
* neuropathy
* chronic narcotic use
* allergy to local anesthetic solution or NSAIDS
* inability to give consent or cooperate with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Ability to ambulate post operatively. | Up to 3 days (72 hours) post surgery.
  Ability to ambulate and perform tasks of the rehabilitation program and reach rehabilitation milestones after total knee arthroplasty.

SECONDARY OUTCOMES:
Pain scores at rest and with knee flexion. | Up to 3 days ( 72 hours) after surgery
  Measures of pain score using numeric pain rating scale (0=no pain, 10=worst pain) completed by patient in recovery room and every 6 hours for a 72 hour period after discharge from recovery room.
Pain Medication Consumption | Up to 3 days (72 hours) post surgery
  Amount of opioid consumption post surgery for 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, M.D., Principal Investigator — Saint Francis Hospital
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States